CLINICAL TRIAL: NCT07015762
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Dose of IBI3002 in Patients With Atopic Dermatitis - a Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: A Study to Evaluate the Safety and Tolerability of Multiple Dose of IBI3002 in Patients With Atopic Dermatitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI3002T002
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo 4ml SC (Placebo Comparator): Participants with AD will receive Placebo 4ml SC
  Interventions: Drug: Placebo
- IBI3002 300mg SC (Experimental): Participants with AD will receive IBI3002 300mg SC
  Interventions: Drug: IBI3002
- IBI3002 600mg SC (Experimental): Participants with AD will receive IBI3002 600mg SC
  Interventions: Drug: IBI3002
- Placebo 2ml SC (Placebo Comparator): Participants with AD will receive Placebo 2ml SC
  Interventions: Drug: Placebo
- Placebo 1ml SC (Placebo Comparator): Participants with AD will receive Placebo 1ml SC
  Interventions: Drug: Placebo
- IBI3002 150mg SC (Experimental): Participants with AD will receive IBI3002 150mg SC
  Interventions: Drug: IBI3002

INTERVENTIONS:
Drug: IBI3002 — Participants with AD will receive IBI3002 at the corresponding dose and dosing interval.
  Arms: IBI3002 150mg SC; IBI3002 300mg SC; IBI3002 600mg SC
Drug: Placebo — Participants with AD will receive placebo at the corresponding volume and dosing interval.
  Arms: Placebo 1ml SC; Placebo 2ml SC; Placebo 4ml SC

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study aimed at evaluating the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of IBI3002 in participants with moderate to severe atopic dermatitis (AD). The study plans to enroll patients with moderate to severe AD who have a poor response to topical treatment or who are not suitable for topical treatments. It aims to evaluate the safety, tolerability, PK characteristics, immunogenicity, PD characteristics, and changes in clinical characteristics of these participants receiving multiple doses of IBI3002.

The entire study includes the screening period (4 weeks before dosing), the dosing period (12 weeks), and the safety follow-up period (8 weeks).

The study plans to enroll 9 to 27 participants with moderate to severe AD, who will be randomly assigned in a 1:1:1 ratio to the following 3 cohorts to receive subcutaneous injection of the corresponding dose of IBI3002 or a matching volume of placebo. Investigators and participants remain blind within the same cohort.

Cohort 1: 150mg SC (IBI3002: placebo=2 :1); Cohort 2: 300mg SC (IBI3002: placebo=2 :1); Cohort 3: 600mg SC( IBI3002: placebo=2 :1);

The participants need to be observed at the study site for 3 hours after each dose and are allowed to leave after investigators determine no safety risk.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years.
2. Weight ≥40kg.
3. Meet the diagnostic criteria of the Hannifin & Rajka criteria, and have been diagnosed with AD for ≥12 months at screening. If determined by Investigators, previous diagnostic terms like "dermatitis" and "eczema" are also acceptable.
4. Have an Eczema area and severity index (EASI) score ≥16, the Investigator´s Global Assessment score ≥3, and the involved Body Surface Area (BSA) ≥10% at screening and randomization.

Exclusion Criteria:

1. Having any disease that have an impact on the participant's own safety or participation in the study. Including but not limited to mental disorders, diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system or metabolic system, in the opinion of Investigator.
2. Participants with a known history of active tuberculosis or clinically suspected manifestations of tuberculosis (including but not limited to pulmonary tuberculosis, lymph node tuberculosis, tuberculous pleurisy, etc.); Or chest imaging suggests the existence of suspected evidence of tuberculosis; Or there is any other clinical evidence of latent tuberculosis. Those with positive T-SPOT.TB need to receive preventive anti-tuberculosis treatment from 4 weeks before the first dose until the end of the study. If the participant is judged by Investigator to be intolerant to preventive anti-tuberculosis treatment, they should not be included in the study either.
3. A history of malignant tumors, except for resected or cured localized basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin.
4. The peripheral blood white blood cells or neutrophils are lower than the lower limit of the normal value, at screening or randomization.
5. The co-existing of any other skin comorbidities that may interfere with the assessment related to AD, in the opinion of Investigators.

The above information is not intended to contain all considerations relevant to a participant's potential participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple doses of IBI3002 in Atopic Dermatitis patients. | Baseline to Week 20
  The incidence of Adverse events (AE) and Serious Adverse events (SAE) in participants with AD after multiple doses of IBI3002;

SECONDARY OUTCOMES:
To evaluate the PK parameters of IBI3002 in participants with AD; | Baseline to Week 20
  PK parameters include, the maximum concentration (Cmax), after multiple doses.
To evaluate the PK parameters of IBI3002 in participants with AD; | Baseline to Week 20
  PK parameters include, the maximum concentration (Tmax), after multiple doses.
To evaluate the PK parameters of IBI3002 in participants with AD; | Baseline to Week 20
  PK parameters include, the maximum concentration (AUC), after multiple doses.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China